CLINICAL TRIAL: NCT03870685
Title: Surgical Site Infiltration of Liposomal Bupivacaine Versus Transversus Plane Block With Liposomal Bupivacaine in Patients With Suspected or Known Gynecologic Cancer Undergoing Laparotomy Via Midline Incision
Brief Title: Surgical Site Infiltration of Exparel vs TAP Block With Exparel in Patients Undergoing Laparotomy Via Midline Incision
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danbury Hospital (Other)
Responsible Party: Principal Investigator, Linus Chuang, Network Chairman OB/GYN, Danbury Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-701
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Patients randomized to TAP block with liposomal bupivacaine OR surgical site infiltration of liposomal bupivacaine for postoperative analgesia after undergoing midline laparotomy
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAP block with Exparel (Active Comparator): Patients will receive immediate postoperative bilateral 2-quadrant TAP block with Exparel (liposomal bupivacaine) admixed with bupivacaine HCl and saline by the anesthesia team.
  Interventions: Procedure: TAP Block; Drug: Exparel
- Surgical Site Infiltration of Exparel (Active Comparator): Patients will receive surgical site infiltration of Exparel (liposomal bupivacaine) admixed with bupivacaine HCl and saline by surgeon.
  Interventions: Procedure: Surgical Site Infiltration; Drug: Exparel

INTERVENTIONS:
Procedure: TAP Block — Transversus Plane block
  Arms: TAP block with Exparel
Procedure: Surgical Site Infiltration — Surgical Site Infiltration
  Arms: Surgical Site Infiltration of Exparel
Drug: Exparel — liposomal bupivacaine

SUMMARY:
This is a randomized-controlled prospective study to be conducted at Danbury Hospital and Norwalk Hospital to compare postoperative opioid consumption and pain scores of patients with suspected or known gynecologic malignancies undergoing midline laparotomy who received TAP block with liposomal bupivacaine versus surgical site infiltration of liposomal bupivacaine.

Primary outcome: Total postoperative opioid consumption as measured by morphine equivalents over 48 hour period.

Secondary outcomes include: Pain scores (based on visual analog scale 1-10) at 2 hours, 6 hours, 12 hours, 24 hours and 48 hours postoperatively at rest and upon exertion (Valsalva maneuver), Severity of nausea, Episodes of vomiting, Total antiemetics consumption over 48 hour period.

DETAILED DESCRIPTION:
Recent studies suggest surgical site infiltration of local anesthetic into the preperitoneal, subfascial and/or subcutaneous planes as an alternative approach. The literature suggests this offers superior pain relief and significantly reduced morphine consumption. This procedure has been shown to provide excellent analgesia in open inguinal hernia repair and colorectal procedures up to 72 hours after a single injection. However, there is limited published data comparing TAP block with liposomal bupivacaine and surgical site infiltration of liposomal bupivacaine in open hysterectomy patients.

The investigators propose to prospectively study the efficacy of surgical site infiltration of liposomal bupivacaine versus TAP block with liposomal bupivacaine in patients with suspected or known gynecologic malignancies undergoing midline laparotomy. The investigators hypothesize that surgical site infiltration of liposomal bupivacaine is more effective than TAP block with liposomal bupivacaine in this patient population. The investigators primary outcome will be postoperative total 48 hour opioid consumption.

Secondary outcomes will include visual analog scale (VAS) pain scores at rest and upon exertion (Valsalva maneuver) at 2 hours, 6 hours, 12 hours, 24 hours and 48 hours postoperatively, severity of nausea, episodes of vomiting and total antiemetics consumption postoperatively. Pain scores and severity of nausea scores will be collected in person or over the phone.

The investigators expect the results of this study to demonstrate that surgical site infiltration of liposomal bupivacaine in patients with suspected or known gynecologic malignancies undergoing midline laparotomy may help shorten the recovery period and reduce the need for postoperative opioid medications. Furthermore, generally patients undergoing procedures such as tumor debulking and lymph node dissection would have an extended hospitalization. If surgical site infiltration of liposomal bupivacaine administration is found to decrease the length of hospitalization (versus TAP Block with liposomal bupivacaine), it will significantly decrease the health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Any woman age 18 or over with known or suspected gynecologic malignancy who is scheduled for laparotomy via vertical midline incision at Danbury Hospital or Norwalk Hospital
* American Society of Anesthesiologists physical status I to IV (a normal healthy patient to a patient with severe systemic disease that may be constant threat to life)
* English or Spanish speaking

Exclusion Criteria:

* Pregnancy
* Unable to obtain consent
* Severe allergies and/or anaphylaxis to bupivacaine or other anesthetics of the same class, to hydromorphone or morphine equivalents
* Patients taking fospropofol, hyaluronidase, propofol, propranolol, St John's Wort and verapamil at the time of screening
* Significant psychiatric disturbance as recorded in the medical record
* Current or history of alcohol or drug addiction
* Have current acute or chronic pain disorders as indicated in medical record
* Current or history of opioid dependence
* Contraindications to acetaminophen (significant hepatic dysfunction or disease), ketorolac and ibuprofen (significant renal dysfunction or reactive airway disease)
* ≥2 previous midline laparotomies
* BMI >45

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Total postoperative opioid consumption over 48 hours | over 48 hour period after surgery
  Total postoperative opioid consumption as measured by morphine milligram equivalents (MME)

SECONDARY OUTCOMES:
Pain scores at rest and upon exertion | 2 hours, 6 hours, 12 hours, 24 hours and 48 hours postoperatively
  Pain scores based on Wong-baker FACES Pain Rating Scale (Visual analog scale (VAS)) at rest and upon exertion (Valsalva maneuver) will be collected in person or over the phone. 0 - no hurt, 2 - hurts little bit, 4 - hurts little more, 6 - hurts even more, 8 - hurts whole lot, 10 - hurts worst.
Severity of nausea | 2, 6, 12, 24, & 48 hours postoperatively
  Severity of nausea will be collected in person or over the phone. Severity of Nausea Scale:- 0 = none, 1 = mild, 2 = moderate, 3 = severe
Episodes of vomiting | 48 hours postoperatively
  Total number of vomiting episodes will be collected from medical record.
Total antiemetics consumption | 48 hour postoperatively
  Total antiemetics consumption (type of antiemetic, mode of administration, dose, time of administration) will be collected from medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Linus Chuang, MD, Principal Investigator — Danbury Hospital, Nuvance Health
Locations (1):
- Danbury Hospital, Danbury, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atim A, Bilgin F, Kilickaya O, Purtuloglu T, Alanbay I, Orhan ME, Kurt E. The efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing hysterectomy. Anaesth Intensive Care. 2011 Jul;39(4):630-4. doi: 10.1177/0310057X1103900415. PMID 21823381
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] Abdallah FW, Halpern SH, Margarido CB. Transversus abdominis plane block for postoperative analgesia after Caesarean delivery performed under spinal anaesthesia? A systematic review and meta-analysis. Br J Anaesth. 2012 Nov;109(5):679-87. doi: 10.1093/bja/aes279. Epub 2012 Aug 19. PMID 22907337
- [Background] Brogi E, Kazan R, Cyr S, Giunta F, Hemmerling TM. Transversus abdominal plane block for postoperative analgesia: a systematic review and meta-analysis of randomized-controlled trials. Can J Anaesth. 2016 Oct;63(10):1184-1196. doi: 10.1007/s12630-016-0679-x. Epub 2016 Jun 15. PMID 27307177
- [Background] Joshi GP, Rawal N, Kehlet H; PROSPECT collaboration; Bonnet F, Camu F, Fischer HB, Neugebauer EA, Schug SA, Simanski CJ. Evidence-based management of postoperative pain in adults undergoing open inguinal hernia surgery. Br J Surg. 2012 Feb;99(2):168-85. doi: 10.1002/bjs.7660. Epub 2011 Sep 16. PMID 21928388
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Hotta K, Inoue S, Taira K, Sata N, Tamai K, Takeuchi M. Comparison of the analgesic effect between continuous wound infiltration and single-injection transversus abdominis plane block after gynecologic laparotomy. J Anesth. 2016 Feb;30(1):31-8. doi: 10.1007/s00540-015-2083-z. Epub 2015 Oct 14. PMID 26467038
- [Background] Gasanova I, Alexander J, Ogunnaike B, Hamid C, Rogers D, Minhajuddin A, Joshi GP. Transversus Abdominis Plane Block Versus Surgical Site Infiltration for Pain Management After Open Total Abdominal Hysterectomy. Anesth Analg. 2015 Nov;121(5):1383-8. doi: 10.1213/ANE.0000000000000909. PMID 26252171